CLINICAL TRIAL: NCT00099463
Title: A Phase I Study of the Safety and Immunogenicity of a SARS Recombinant DNA Plasmid Vaccine, VRC-SRSDNA015-00-VP, in Healthy Adult Volunteers
Brief Title: Phase I Study of a Vaccine for Severe Acute Respiratory Syndrome (SARS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050056; 05-I-0056
Record Dates: First submitted 2004-12-14; First posted 2004-12-15 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-08-22

CONDITIONS: Healthy
Keywords: Coronavirus; Healthy; Immunity; Preventive; Virus; Healthy Volunteer; HV
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases | interventions — Hematologic Tests; Urinalysis; Restraint, Physical; Vaccines

INTERVENTIONS:
Procedure: Blood Test
Procedure: Urine Test
Procedure: Physical Exam
Drug: Vaccine
Drug: VRC-SRSDNA015-00-VP

SUMMARY:
This study will test whether an experimental vaccine to protect against severe acute respiratory syndrome (SARS) is safe, causes any side effects, and causes an immune response. SARS affects the respiratory system, usually starting with fever and muscle aches. Patients may get a dry cough and have difficulty breathing. Infection may be mild, but it can lead to death.

Vaccines contain substances from an infectious agent, such as a virus, that, when injected into a person's body, stimulates production of antibodies that create resistance, or immunity, to that agent. The vaccine in this study contains genetic material (DNA) that codes for a protein found in the virus that causes SARS. Injected into a muscle, it instructs the body to make a small amount of a SARS protein. The vaccine is made from just one small part of the code for one SARS protein; a person cannot get SARS from the vaccine.

Normal volunteers between 18 and 50 years of age who are in general good health may be eligible for this 32-week study. Candidates are screened with a physical examination and blood and urine tests.

Participants have nine clinic visits during the study. They receive three vaccine injections, given with a system called the Bioinjector 2000® (Registered Trademark), which delivers the vaccine through the skin without the use of a needle. Following each injection, participants take home a diary card, on which they record their temperature and any vaccine side effects daily for 5 days. Participants must immediately report any symptoms to a study physician, and, if necessary, go to the clinic for an examination. Participants have the following tests and procedures:

* Vaccine injections (study day 0, around week 4, and around week 8, with at least 21 days between injections)
* Medical history and, if needed, physical examination (study day 0 and weeks 2, 4, 6, 8, 10, 12, 24, and 32)
* Check of vital signs and weight (study day 0 and weeks 2, 4, 6, 8, 10, 12, 24 and 32)
* Lymph node examination (day 0 and weeks 2, 4, 6, 8, 10 and 12)
* Blood draw (study day 0 and weeks 2, 4, 6, 8, 10, 12, 24 and 32)
* Pregnancy test for women (day 0 and weeks 4, 8 and 32)
* Urine sample (day 0 and weeks 2, 4, 6, 8, 10)

DETAILED DESCRIPTION:
Study Design: This is a Phase I open label study to evaluate safety, tolerability, and immune response of a recombinant DNA vaccine, VRC-SRSDNA015-00-VP. The hypothesis is that this regimen will be safe for human administration and elicit immune responses to the SARS coronavirus (CoV) spike (S) protein. The primary objective is to evaluate the safety and tolerability in humans of the investigational vaccine. Secondary and exploratory objectives are related to the immunogenicity of the study vaccine.

Product Description: VRC-SRSDNA015-00-VP is composed of a single closed, circular DNA plasmid that is based on the S protein of SARS-CoV. Vaccine vials will be supplied at 4 mg/mL. Each DNA vaccination will be 1 mL of vaccine administered intramuscularly (in deltoid muscle) using the Biojector 2000 Needle-Free Injection Management System.

Subjects: Healthy adult volunteers (18 to 50 years old) will be enrolled.

Study Plan: Ten volunteers will be enrolled and receive 3 injections on the schedule shown in the schema. The protocol requires nine clinic visits and three telephone follow-up contacts.

Study Duration: 32 weeks clinical follow-up for each participant.

Study Endpoints: The primary endpoint is safety of the regimen; secondary immunogenicity endpoints are an intracellular cytokine staining (ICS) assay for SARS specific T cell responses and an assay for antibody-dependent enhancement of virus uptake. The principal timepoints for ICS are Week 0 (baseline) and Weeks 6, 8, 10 and 12. ICS at other study timepoints, as well as other immunogenicity assays through Week 32, will be completed as exploratory evaluations.

ELIGIBILITY:
* INCLUSION CRITERIA:

A participant must meet all of the following criteria:

18 to 50 years old.

Available for clinical follow-up through Week 32 of the study.

Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.

Complete an Assessment of Understanding prior to enrollment and verbalize understanding of all questions answered incorrectly.

Able and willing to complete the informed consent process.

Willing to receive HIV test results and wiling to abide by NIH guidelines for partner notification of positive HIV results.

Willing to donate blood for sample storage to be used for future research.

In good general health without clinically significant medical history and has satisfactorily completed screening.

Physical examination and laboratory results without clinically significant findings within the 28 days prior to enrollment.

Laboratory Criteria within 28 Days prior to Enrollment:

Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to 13.5 g/dL for men.

WBC = 3,300-12,000 cells/mm(3).

Absolute neutrophil count (ANC) within institutional normal range.

Total lymphocyte count greater than or equal to 800 cells/mm(3).

Platelets within institutional normal limits.

ALT (SGPT) less than or equal to upper limit of normal.

Serum creatinine less than or equal to upper limit of normal.

Normal urinalysis defined as negative glucose, negative or trace protein, and no clinically significant blood in the urine.

Negative FDA-approved HIV blood test. (Note: Results of HIV ELISA will be documented, but a negative HIV PCR will be sufficient for eligibility screening of subjects with positive HIV ELISA that is due to prior participation in an HIV vaccine study).

Negative Hepatitis B surface antigen.

Negative anti-HCV (hepatitis C virus antibody) and negative HCV PCR.

Female Specific Criteria:

Negative beta-HCG pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential.

A female participant must meet any of the following criteria:

No reproductive potential because of menopause [one year without menses] or because of a hysterectomy, bilateral oophorectomy, or tubal ligation;

Or

Participant agrees to be heterosexually inactive at least 21 days prior to enrollment and through Week 32 of the study;

Or

Participant agrees to consistently practice contraception at least 21 days prior to enrollment and through Week 32 of the study by one of the following methods:

Condoms, male or female, with or without a spermicide;

Diaphragm or cervical cap with spermicide;

Intrauterine device;

Contraceptive pills or patch, Norplant, Depo-Provera or other FDA-approved contraceptive method;

Male partner has previously undergone a vasectomy for which there is documentation.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

Women:

Woman who is breast-feeding or planning to become pregnant during the 32 weeks of study participation.

Volunteer has received any of the following substances:

Immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis).

Blood products within 120 days prior to HIV screening.

Immunoglobulin within 60 days prior to HIV screening.

Investigational research agents within 30 days prior to initial study vaccine administration.

Live attenuated vaccines within 30 days prior to initial study vaccine administration.

Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days of study vaccine administration.

Current anti-TB prophylaxis or therapy.

Volunteer has a history of any of the following clinically significant conditions:

Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain.

Autoimmune disease or immunodeficiency.

Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.

Diabetes mellitus (type I or II), with the exception of gestational diabetes.

History of thyroidectomy or thyroid disease that required medication within the past 12 months.

Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years.

Hypertension that is not well controlled by medication or is more than 145/95 at enrollment.

Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.

Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of study.

Seizure disorder other than: 1) febrile seizures under the age of two, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure not requiring treatment within the last 3 years.

Asplenia, functional asplenia or any condition resulting in the absence or removal o the spleen.

Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years; disorder requiring lithium; or suicidal ideation occurring within five years prior to enrollment.

Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Allergic reaction to aminoglycoside antibiotics.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10
Dates: Start 2004-12-09; Study Completion 2007-08-22

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ksiazek TG, Erdman D, Goldsmith CS, Zaki SR, Peret T, Emery S, Tong S, Urbani C, Comer JA, Lim W, Rollin PE, Dowell SF, Ling AE, Humphrey CD, Shieh WJ, Guarner J, Paddock CD, Rota P, Fields B, DeRisi J, Yang JY, Cox N, Hughes JM, LeDuc JW, Bellini WJ, Anderson LJ; SARS Working Group. A novel coronavirus associated with severe acute respiratory syndrome. N Engl J Med. 2003 May 15;348(20):1953-66. doi: 10.1056/NEJMoa030781. Epub 2003 Apr 10. PMID 12690092